CLINICAL TRIAL: NCT04653012
Title: Multi-level Approach of Brain Activity Using Intracranial Electrodes in Epileptic Patients
Acronym: EpiMicro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C19-55; 2020-A00445-34 (Registry Identifier: ID RCB)
Record Dates: First submitted 2020-11-05; First posted 2020-12-04 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Focal Epilepsy; Electrodes, Implanted; Cognitive Function; Neurophysiology
Keywords: Microelectrodes; Seizures; EEG
MeSH Terms: conditions — Epilepsies, Partial; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Macro-microelectrode implantation (Experimental): Implantation of macro-micro electrodes of the Adtech Benkhe-Fried type in epileptic patients who are undergoing evaluation with intracranial EEG electrodes
  Interventions: Device: Intracranial macro-microelectrode recording

INTERVENTIONS:
Device: Intracranial macro-microelectrode recording — Additionnally to clinical macroelectrodes, Benkhe-Fried depth macro-microelectrodes will be implanted and recorded during the pre-surgical investigation of epileptic patients

SUMMARY:
The main goal of this project is to study the mechanisms of epileptic activities using intracranial macro and micro electrodes in epileptic patients undergoing pre-surgical investigation.

The recordings will also be used to study physiological mechanisms like sleep and different cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with focal drug-resistant epilepsy
* Patients who undergo a presurgical evaluation with intracranial electrodes in the videoEEG unit of the Neurology department at the Pitié-Salpêtrière hospital.
* Patients who have been informed and provided written informed consent to take part in the study

Exclusion Criteria:

* Contraindication for an intracranial investigation (with macro-electrodes) : intercurrent infectious syndrome, decompensated associated pathology (cardiac, pulmonary, renal, hepatic), patient with increased risk of infection (ex: under immunosuppressive therapy)
* Pregnant or parturient woman
* Breastfeeding woman
* Minor person or legally protected adult (tutelage, legal guardianship, maintenance of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-28 (Actual); Primary Completion 2029-02-27 (Estimated); Study Completion 2031-02-27 (Estimated)

PRIMARY OUTCOMES:
Identification of single unit changes at seizure emergence | Whole duration of the clinical inverstigation, until 4 weeks
  In order to identify biomarkers of epileptic seizures we will study single neuron activities (firing rate) using spike sorting at different time periods (before, during and after seizures and during interictal periods)
  We expect to observe significant changes in firing rate across the different time periods.
Identification of local field potential (LFP) changes at seizure emergence | Whole duration of the clinical inverstigation, until 4 weeks
  In order to identify biomarkers of epileptic seizures we will study LFP power using time frequency analysis at different time periods (before, during and after seizures and during interictal periods)
  We expect to observe significant changes in LFP power across the different time periods.

SECONDARY OUTCOMES:
Comparison of single unit activity before seizure according to brain localization | Whole duration ofthe clinical inverstigation, until 4 weeks
  We will compare firing rate before seizure according to brain regions (anatomy and involvement in the seizure onset zone)
Identification of single unit changes during physiological brain activity | Whole duration ofthe clinical inverstigation, until 4 weeks
  We will compare firing rates during resting states and stimulus induced states.
  We expect to observe significant changes in firing rate between states.
Identification of LFP power changes during physiological brain activity | Whole duration ofthe clinical inverstigation, until 4 weeks
  We will compare LFP power during resting states and stimulus induced states.
  We expect to observe significant changes in LFP power between states.
Multilevel study of brain activity | Whole duration ofthe clinical inverstigation, until 4 weeks
  We will look for correlation between firing rates and LFP power changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No